CLINICAL TRIAL: NCT05408858
Title: LGBTQ-affirmative Cognitive Behavioral Group Therapy for Youth: A Pilot Study
Brief Title: LGBTQ-affirmative CBT for Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000030664
Record Dates: First submitted 2022-05-19; First posted 2022-06-07 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2023-12

CONDITIONS: Anxiety Disorders; Depression; LGBTQ
Keywords: minority stress; LGBTQ
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LGBTQ-affirmative cognitive behavioral group therapy (Experimental): LGBTQ-affirmative cognitive behavioral group therapy consists of 10 weekly, 90-minute group therapy sessions, delivered remotely via Zoom. Intervention sessions and associated home practice will cover the following topics: Building and keeping motivation; Introduction to LGBTQ-related stress; Getting to know your emotions; Introduction to emotional behaviors and behavioral experiments; Awareness of physical sensations and introduction to flexible thinking; Being flexible in your thinking; Awareness of emotional experiences; Assertiveness; Situational exposures; Reviewing accomplishments and looking ahead. Participants will be taught intervention content through a range of teaching modalities including use of the Zoom whiteboard feature, videos, interactive activities, worksheets, and group discussion.
  Interventions: Behavioral: LGBTQ-affirmative cognitive behavioral group therapy

INTERVENTIONS:
Behavioral: LGBTQ-affirmative cognitive behavioral group therapy — 10 sessions of supportive, LGBTQ-affirmative psychotherapy

SUMMARY:
This study will adapt LGBTQ-affirmative cognitive behavior therapy (CBT) - previously only used with adults - for youth aged 12-17 years. This intervention addresses the pathways through which minority stress compromises lesbian, gay, bisexual, transgender, and queer (LGBTQ) young peoples' mental health. The purpose of this study is to determine if the intervention is acceptable and feasible for LGBTQ youth.

DETAILED DESCRIPTION:
Lesbian, gay, bisexual, transgender, and queer (LGBTQ) youth experience more mental health problems than their heterosexual and cisgender peers. The purpose of the proposed mixed-methods study is to assess the feasibility, acceptability, and need for refinement of LGBTQ-affirmative cognitive behavior therapy for youth aged 12-17 years in New York, New Jersey, and Connecticut. This study will be the first to adapt the randomized controlled trial tested LGBTQ-affirmative CBT intervention for youth, and the first to deliver it in a virtual group format. Qualitatively, investigators will conduct structured post-treatment interviews to assess the feasibility, acceptability, and refinement of the intervention in this population. Quantitatively, investigators will assess the feasibility and acceptability of the intervention through analysis of indices like number of sessions attended, number of homework assignments completed, weekly treatment satisfaction ratings, and a post-treatment feedback survey. Investigators will also examine changes from pre- to post-treatment in youth's mental health symptoms, minority stress reactions, and emotional regulation and coping difficulties. These pilot data will be used to estimate the sample sizes needed for a future, larger trial of this treatment, as well as areas in which the treatment could be refined.

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years old
* Self-identify as LGBTQ (any diverse sexual orientation and/or gender identity)
* Live in New York, New Jersey, or Connecticut
* Fluent in English
* Meet diagnostic criteria for a DSM-5 internalizing disorder (any depressive, anxiety, obsessive-compulsive, or adjustment disorder)
* Have consistent, weekly access to an Internet-enabled electronic device that allows for video-conferencing
* Availability to attend 10 weekly 90 minute intervention sessions in summer 2021
* Access to a quiet, private place for intervention sessions
* Provision of informed consent from parent/guardian and assent from the youth

Exclusion Criteria:

* Evidence of any psychotic or bipolar spectrum diagnosis
* Active suicidality and/or homicidality (defined as active intent or concrete plan, as opposed to passive ideation) or psychiatric hospitalization within the past 6 months
* Significant cognitive impairment (as determined by an intellectual disability screener) or significant developmental disorder (if impairing youth's ability to participate in group therapy)
* Significant behavior disorder (e.g., oppositional defiant disorder, conduct disorder) if impairing youth's ability to participate in group therapy
* Currently in mental health treatment exceeding one day per month
* Received any cognitive-behavioral therapy treatment in the past 12 months
* Unstable psychotropic medications (defined as changes to antidepressant dosage in the past 3 months, or changes to a benzodiazepine dosage in the past month)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Participant identifies as either a gender minority (e.g., transgender, nonbinary) or as a sexual minority (e.g., gay, bisexual)
Enrollment: 9 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pachankis, PhD, Principal Investigator — Yale University
Locations (1):
- Dr. Pachankis' Lab, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 12 months after study completion for three years.
Access Criteria: Data access requests from qualified academic investigators for non-commercial research interests will be reviewed by study investigators. Requestors will be required to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was advertised to potential participants using social media (Facebook and Twitter). Study team also sent emails to LGBTQ organizations in the Tri-state area to promote the study.
Period: Overall Study
Arm/Group | LGBTQ-affirmative Cognitive Behavioral Group Therapy
Started | 9
Completed | 8
Not Completed | 1
Not completed — no longer met eligibility criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | LGBTQ-affirmative Cognitive Behavioral Group Therapy
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.89 (1.36)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Transgender girl | 1
  Cisgender girl | 2
  Transgender boy | 1
  Nonbinary | 3
  Nonbinary/questioning | 1
  Genderfluid | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9
Grade in School [Count of Participants; unit: Participants]
  7th | 1
  8th | 1
  9th | 4
  10th | 2
  11th | 1
Sexual Orientation [Count of Participants; unit: Participants]
  Lesbian | 1
  Bisexual | 3
  Queer | 1
  Asexual | 3
  Panromantic asexual | 1

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction With Treatment
Description: Client satisfaction with treatment will be measured through the Client Satisfaction Questionnaire-8 (CSQ-8; Larsen et al., 1979), a well-validated, 8-item self-report questionnaire designed to assess patient/client satisfaction with services received. Both the adolescent self-report and the parent report of child services versions of the CSQ-8 will be used in this study. Items are scored on a 4-point scale, where higher scores indicate more satisfaction. Total score is determined by summing the 8 items, yielding a score between 8 and 32. The CSQ-8 has demonstrated excellent internal consistency in prior studies (alpha = 0.93)
Time Frame: Immediate Post-treatment at Week 10
Population: Only 8 participants were analyzed, as 1 participant was dismissed after session 2 for not meeting eligibility criteria.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LGBTQ-affirmative Cognitive Behavioral Group Therapy
Number analyzed (Participants) | 8
score on a scale | 27.13 (5.22)

2. Secondary Outcome: Session Attendance
Description: Participant session attendance will be tracked by the study therapist each week to examine the feasibility of weekly sessions. Attendance will be scored as an average of summed weekly attendance counts per participant.
Time Frame: Immediate Post-treatment at Week 10
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | LGBTQ-affirmative Cognitive Behavioral Group Therapy
Number analyzed (Participants) | 9
sessions | 7 (3.04)

ADVERSE EVENTS:
Time Frame: From enrollment to completion of the final follow-up survey, up to 19 weeks.
Arm/Group | LGBTQ-affirmative Cognitive Behavioral Group Therapy
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT05408858/Prot_SAP_000.pdf